CLINICAL TRIAL: NCT04680247
Title: Outcome After Polyaxial Locking Plate Osteosynthesis in Proximal Tibia Fractures: a Prospective Clinical Trial
Brief Title: Polyaxial Locking Plate Osteosynthesis in Proximal Tibia Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dominik Völk, Principal Investigator, Technical University of Munich
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5923/13
Record Dates: First submitted 2020-12-07; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Tibia Plateau Fracture
Keywords: Proximal tibia fracture; clinical trial; polyaxial locking plate; outcome; osteosynthesis
MeSH Terms: conditions — Tibial Plateau Fractures

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VA-LCP (Active Comparator): Osteosynthesis with a VA-LCP system
  Interventions: Procedure: VA-LCP
- NCB-PT (Active Comparator): Osteosynthesis with a NCB-PT system
  Interventions: Procedure: NCB-PT

INTERVENTIONS:
Procedure: VA-LCP — Surgery using the VA-LCP implant
  Arms: VA-LCP
Procedure: NCB-PT — Surgery using the NCB-PT implant
  Arms: NCB-PT

SUMMARY:
From October 2013 28 patients with proximal tibia fractures (AO/ASIF 41 B-C) were included in this study. According to our treatment algorithm for this entity Patients were assigned into two groups and treated with different polyaxial locking plates (NCB-PT®, Zimmer vs. VA-LCP® Synthes). After 12 months postoperative the investigators conducted clinical and radiological follow-ups.

DETAILED DESCRIPTION:
Prior to the onset of the study, the approval by the medical ethics committee of the Technical University of Munich (TUM) (Trial Number: 5923/13) was obtained. During a period from October 2013 to December 2015 the investigators enrolled 28 patients aged 25 to 82 into our study. All patients suffered a fracture of the proximal tibia. The fractures were classified according to the AO/OTA classification. Every one of the 28 patients had an indication for locking plate osteosynthesis. The investigators included all type 41-B fractures and all type 41-C fractures. Pathological fractures, pregnancy, adolescence (age <18 y), prisoners and patients currently put under tutelage were excluded. The patients were scheduled for a locking plate osteosynthesis with either the NCB-PT® system or the VA-LCP® system. The discission was made by using our internal treatment algorithm for proximal tibia fractures. Age, bone quality, fracture configuration, allergies and distal fracture extension were among the criteria the investigators took into account to determine the plate type.

Surgical technique

The surgical technique was standardized, as far as possible. All surgeons agreed upon the following procedure. The anterolateral approach was used in all cases. Depending on the fracture type and the damaged column the standard approach was supplemented with either a posterolateral approach or a posteromedial approach. After arthrotomy and suturing of the lateral meniscus the fracture was reduced. This was performed under direct visual control of the joint surface and/or image intensifier. K-wires and/or a reduction forceps was used to secure the reduction. Afterwards the locking plate was inserted and temporarily fixed to the bone with K-wires. After checking the correct position of the plate with an image intensifier the screws were applied. In case of VA-LCP®, additional lag screws have been inserted at discretion of the surgeon. All patients received a perioperative single shot antibiotics. Our postoperative procedure consisted of a partial weight bearing for 6 weeks for all patients. Regarding the allowed range of motion the investigators distinguished two different groups: patient who received an arthrotomy and a refixation of the meniscus ought to comply with a limited range of motion for 6 weeks overall (week 1-2 30/0/0, week 3-4 60/0/0, week 5-6 90/0/0, week 7 free RoM). Patients with no arthrotomy were allowed free range of motion immediately after surgery.

Postoperative clinical and radiologic follow-up The investigators conducted the follow up after 12 months. The clinical evaluation was performed in our trauma outpatient clinic. With the help of standardized questionnaires, the investigators examined amongst others: the range of motion, cruciate ligament/ collateral ligament instability and meniscus signs to measure the clinical outcome. Also the investigators collected data from 5 different knee scoring systems, the Tegner score, the Rasmussen score (clinical part), the Oxford knee score the Munich knee questionnaire and the Lysholm score. To measure the patient satisfaction the investigators used the SF36 (36-Item Short-Form Health Survey) Besides the clinical data the primary outcome measurements also included standardized, blinded radiological evaluation. The investigators conducted X-ray examinations in two plains (AP, lateral view) and examined them for signs of screw misplacement, primary/secondary loss of reduction, non-union and malalignment.

Statistics The statistical analysis was performed with the program GraphPad Prism 6 (GraphPad Software Inc., La Jolla, CA, USA). To check the data for standard distribution the investigators used the D'Agostino omnibus K2 test. For continuous parametric variables the investigators used the Student's t-test, for non-parametric variables the Mann-Whitney U test and for binominal variables the Fisher's exact test. In all analysis the significance level was set at a p-value <0,05, the investigators plotted the data as mean values ± SEM.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 25 to 82 with a proximal tibia fractures (AO/ OTA 41 B-C) and indication for locking plate osteosynthesis

Exclusion Criteria:

* Pathological fractures
* pregnancy
* adolescence (age <18 y)
* prisoners
* patients currently put under tutelage

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10-05 (Actual); Primary Completion 2016-12-14 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Rasmussen score | 12 months
  functionality and pain
Tegner score | 12 months
  activity, functionality
Rasmussen score (radiological part) | 12 months
  articular surface depression, condylar widening and fragment angulation
Fracture healing | 12 months
  Categorized in accordance to the phases of bone healing: A = cloudy cortical edges and condensation (granulation phase), B = defined edges bridging, lamellar bone deposition, cartilage callus formation (reparative phase), C = remodelling to original bone contour (remodelling phase), D = non-union
Lysholm score | 12 months
  functionality and pain
Oxford knee score | 12 months
  functionality and pain
Munich knee questionnaire | 12 months
  pain, daily life and sports activity, functionality

CONTACTS AND LOCATIONS:
Overall Officials: Peter Biberthaler, Prof, Study Director — Technical University of Munich Klinikum rechts der Isar, Department of Trauma Surgery; Marc Hanschen, PD, Study Chair — Technical University of Munich Klinikum rechts der Isar, Department of Trauma Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Volk D, Neumaier M, Einhellig H, Biberthaler P, Hanschen M. Outcome after polyaxial locking plate osteosynthesis in proximal tibia fractures: a prospective clinical trial. BMC Musculoskelet Disord. 2021 Mar 18;22(1):286. doi: 10.1186/s12891-021-04158-z. PMID 33736638